CLINICAL TRIAL: NCT03870646
Title: Nebulized hypErtonic Saline for Better Prevention of mUcus pLug in Critical Adult Tracheostomized Patients (the NEBULA Study). A Pilot Randomized Controlled Trial
Brief Title: Nebulized hypErtonic Saline for Better Prevention of mUcus pLug in Critical Adult Tracheostomized Patients
Acronym: NEBULA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Juan Alfonso Soler Barnés, Principal Investigator, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018-11-1-HCUVA
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Critical Illness; Tracheostomy Complication; Mechanical Ventilation Complication; Plug; Mucus
Keywords: Critical Illness; Tracheostomy; Mechanical Ventilation; Complication; Plug; Mucus
MeSH Terms: conditions — Critical Illness | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Unicentre, randomized, two arm, double-blind, controlled trial.
Who Masked: Participant, Care Provider
Masking Description: Identical vials for the intervention and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hypertonic saline (Experimental): Nebulized hypertonic saline of NaCl (7%) in combination with hyaluronic acid
  Interventions: Combination Product: Hypertonic saline of NaCl (7%) in combination with hyaluronic acid
- Isotonic saline (Placebo Comparator): Nebulized isotonic saline of NaCl (0,9%)
  Interventions: Combination Product: Isotonic saline of NaCl (0,9%)

INTERVENTIONS:
Combination Product: Hypertonic saline of NaCl (7%) in combination with hyaluronic acid — Critical adult tracheostomized patients will receive, in the intervention arm, nebulized Hypertonic saline of NaCl (7%) in combination with hyaluronic acid 5ml twice daily for 10 days from the day of the tracheotomy or until decannulation or discharge from the ICU if it happens before. The treatment will be applied through a jet nebulizer located in the inspiratory branch in patients under mechanical ventilation and in the sole tubulant of patients under T-piece oxygen regimen. Salbutamol 100 micrograms / dose, suspension for inhalation in pressure pack: 2 inhalations through the tracheostomy cannula 10 minutes before the application of the nebulization with hypersaline in order to avoid bronchospasm.
  Arms: Hypertonic saline
Combination Product: Isotonic saline of NaCl (0,9%) — Critical adult tracheostomized patients will receive, in the control arm, nebulized isotonic saline of NaCl (0,9%) 5ml twice daily for 10 days from the day of the tracheotomy or until decannulation or discharge from the ICU if it happens before. The treatment will be applied through a jet nebulizer located in the inspiratory branch in patients under mechanical ventilation and in the sole tubulant of patients under T-piece oxygen regimen. Salbutamol 100 micrograms / dose, suspension for inhalation in pressure pack: 2 inhalations through the tracheostomy cannula 10 minutes before the application of the nebulization with isotonic saline in order to avoid bronchospasm.
  Arms: Isotonic saline

SUMMARY:
Tracheostomy is an important tool in the management of respiratory failure in the critically ill patient under mechanical ventilation. Although mechanical ventilation can be a lifesaving intervention, it is also known to carry several side-effects and risks. Among the most frequent complications of mechanical ventilation, obstruction of the airway secondary to a mucus plug is both life threatening and a prevalent phenomenon related to mucociliary system dysfunction, artificial airway itself and the loss of strength that prevents adequate airway clearance. The main indication of tracheostomy is the need for prolonged mechanical ventilation that usually occurs in more severe patients, this circumstance having also been related to the development of intensive care unit (ICU) acquired weakness. Currently, the approach to secretion clearance in critical patients is focused on rehabilitation therapy and humidification. Hypertonic saline (HS) is largely used in cystic fibrosis to increase airways clearance while little evidence is available in other settings although promising results have been reported. In this sense, the use of HS could be beneficial in the prevention of airway obstruction in tracheostomized critical patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Respiratory support through tracheostomy performed during ICU stay.
* Informed consent signed by the relatives or legal representative of the patient.

Exclusion Criteria:

* Pregnancy.
* Any terminal disease.
* Known hypersensitivity to any component of Hyaneb (Hypertonic saline of NaCl (7%) in combination with hyaluronic acid).
* Participation in another research study.
* Any other condition that, according to the investigator, may prevent a participant to complete all the procedures required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with mucus plug | 10 days from the day of the tracheotomy or until decannulation or discharge from the ICU if it happens before.
  Mucus plug will be considered when there is a deterioration of the respiratory support accompanied by at least one of the following:
  * An inability to pass the aspiration catheter through the orotracheal tube or the tracheostomy tube.
  * Sudden hypoxia with physical and / or radiological examination compatible with atelectasis.
  * Need for urgent bronchoscopy with direct vision of the mucous plug.

SECONDARY OUTCOMES:
Length of mechanical ventilation | From the start date of mechanical ventilation to the date of its withdrawal or date of death from any cause, whichever came first, assessed up to 12 months
  Number of days under mechanical ventilation
Percentage of patients died during ICU stay | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 12 months
  Percentage of patients died during ICU stay
Percentage of patients died during hospital stay | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 15 month
  Percentage of patients died during hospital stay
ICU length of stay | From date of ICU admission until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 12 month
  Number of days admitted to the ICU
Hospital length of stay | From date of hospital admission until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 15 month
  Number of days admitted to the hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided